CLINICAL TRIAL: NCT07314645
Title: Strategic Daytime Napping Enhances Agility and Lowers Perceived Exertion But Does Not Improve Fatigue Resistance in Adolescent Soccer Players
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uludag University (Other)
Collaborators: Inonu University (Other); Princess Nourah Bint Abdulrahman University (Other)
Responsible Party: Principal Investigator, Mertkan Öncü, Research Assistant, Uludag University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 2024/5635
Record Dates: First submitted 2025-11-21; First posted 2026-01-02 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Sleep Deprivation; Athletic Performance; Fatigue
Keywords: Daytime Napping; Sleep Inertia; Perceived Exertion; Mood State; Agility; Repeated Sprint Ability; Chronotype
MeSH Terms: conditions — Sleep Deprivation; Fatigue; Idiopathic Hypersomnia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- No Nap (Experimental): No Nap Conditions
  Interventions: Behavioral: Pro Agility Test; Behavioral: Repeated-Sprint Ability (RSA) Test; Behavioral: Rate of Perceived Exertion (RPE)
- 25 Min Nap (Experimental): 25 Min Nap Conditions
  Interventions: Behavioral: Pro Agility Test; Behavioral: Repeated-Sprint Ability (RSA) Test; Behavioral: Rate of Perceived Exertion (RPE)
- 45 Min Nap (Experimental): 45 Min Nap Conditions
  Interventions: Behavioral: Pro Agility Test; Behavioral: Repeated-Sprint Ability (RSA) Test; Behavioral: Rate of Perceived Exertion (RPE)

INTERVENTIONS:
Behavioral: Pro Agility Test — The Pro Agility Test (20-yard shuttle run) evaluates change-of-direction speed. Participants started from the center point, ran 5 yards to the left, then 10 yards to the right, and finally 5 yards back to the center. The total distance was 18.28 meters, and the time to complete the sequence was recorded. Agility and RSA timings were recorded using a dual-beam electronic timing system (SmarTracks, Germany) with a sampling frequency of 1,000 Hz, positioned at the start and finish lines at hip level. This minimized human error and ensured millisecond precision.
Behavioral: Repeated-Sprint Ability (RSA) Test — The RSA test measures an athlete's ability to repeatedly produce maximal sprint efforts with limited recovery. This study employed 6 × 30-meter sprints with 20-second rest intervals between each sprint, a protocol commonly used in team sports to assess anaerobic endurance.
Behavioral: Rate of Perceived Exertion (RPE) — RPE was assessed using the Borg Scale (6-20), which captures the participant's subjective effort during physical activity. RPE was recorded immediately after each sprint during the RSA Test, and the average RPE score represented overall perceived exertion for the session.

SUMMARY:
Background

Daytime napping is increasingly incorporated into athletic recovery routines to manage sleepiness and support alertness. However, the effects of different nap durations on high-intensity anaerobic performance tasks remain insufficiently characterized, particularly in team-sport settings. Nap duration and circadian timing may influence psychomotor readiness, perceived exertion, and fatigue-related responses, yet existing evidence is limited and inconsistent in adolescent athlete populations. This study is designed to examine the acute effects of two daytime nap durations within a controlled experimental framework.

Methods

This study will employ a randomized, crossover design involving sixteen competitive male adolescent soccer players classified as intermediate chronotypes. Each participant will complete three experimental conditions in a randomized order: no nap (N0), a 25-minute nap (N25), and a 45-minute nap (N45), with standardized washout periods between sessions. Nap compliance will be objectively monitored using wrist-worn actigraphy.

Following each condition, participants will observe a standardized 60-minute post-nap wakefulness period prior to performance testing. Agility performance will be assessed using the Pro Agility Test, and anaerobic endurance will be evaluated using a repeated-sprint ability (RSA) protocol. Psychophysiological measures will include ratings of perceived exertion (RPE), the Hooper Index, visual analogue scales (VAS) for subjective alertness, and mood states assessed via the Profile of Mood States (POMS). These outcomes will be collected to compare responses across nap conditions.

Objectives

The primary objective of this study is to compare the acute effects of two daytime nap durations (25 minutes vs 45 minutes) on agility performance in adolescent soccer players without a habitual napping routine. Secondary objectives include examining nap-related differences in repeated-sprint performance indices, perceived exertion, subjective alertness, and mood states.

Keywords

daytime nap; athletic recovery; agility; repeated-sprint ability; perceived exertion; mood; chronotype

ELIGIBILITY:
Inclusion Criteria:

* being a member of the Yeni Malatyaspor U19 or U17 team
* having no history of illness or injury
* no regular napping habit

Exclusion Criteria:

* active infections
* hyperactivity
* sleep disorders
* sleep problems on protocol days

Ages: 16 Years to 19 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes
Enrollment: 16 (Actual)
Dates: Start 2024-05-10 (Actual); Primary Completion 2024-05-18 (Actual); Study Completion 2024-05-18 (Actual)

PRIMARY OUTCOMES:
Pro Agility Test | Immediately after completion of each experimental condition, within a single testing session.
  Change-of-direction performance assessed using the Pro Agility Test (20-yard shuttle run).
  Participants will complete the test following each experimental condition (no nap, 25-minute nap, and 45-minute nap).
  The total time to complete the test will be recorded in seconds using an electronic timing system.
Best sprint (s) | During each experimental testing session, immediately following the nap or no-nap condition.
  Best sprint time measured during a repeated-sprint ability (RSA) test. Participants will perform a standardized RSA protocol consisting of repeated maximal sprints with fixed recovery intervals.
  The fastest single sprint time achieved during each RSA test will be recorded in seconds for each experimental condition (no nap, 25-minute nap, and 45-minute nap) using an electronic timing system.
Total sprint (s) | During each experimental testing session, immediately following the nap or no-nap condition.
  Total sprint time measured during a repeated-sprint ability (RSA) test. Participants will perform a standardized RSA protocol consisting of repeated maximal sprints separated by fixed recovery intervals.
  Total sprint time will be calculated as the sum of all sprint times completed during the RSA test for each experimental condition (no nap, 25-minute nap, and 45-minute nap) and recorded in seconds using an electronic timing system.
4. Rate of Perceived Exertipon (RPE) | Immediately after completion of the repeated-sprint ability test in each experimental session.
  Perceived exertion assessed using the Borg 6-20 Rating of Perceived Exertion (RPE) scale.
  Participants will report their perceived exertion immediately after each sprint during the repeated-sprint ability test.
  The mean RPE score for each testing session will be calculated for each experimental condition.
Hooper Index | After completion of each experimental session, following the nap or no-nap condition.
  Subjective recovery status assessed using the Hooper Questionnaire. The questionnaire evaluates perceived fatigue, stress, muscle soreness, and sleep quality using standardized Likert-scale ratings.
  Participants will complete the Hooper Questionnaire following each experimental condition (no nap, 25-minute nap, and 45-minute nap), and a total Hooper Index score will be calculated for each session.
Subjective Alertness (VAS) | After completion of each experimental session, following the nap or no-nap condition.
  Subjective alertness will be assessed using a visual analogue scale (VAS). Participants will rate their perceived level of alertness on a 100-mm horizontal line anchored by "extremely sleepy" at one end and "fully alert" at the other.
  VAS assessments will be completed following each experimental condition (no nap, 25-minute nap, and 45-minute nap), and the distance from the left anchor will be recorded in millimeters as the alertness score.

SECONDARY OUTCOMES:
Pittsburgh Sleep Quality Index (PSQI) | At baseline, prior to the first experimental session.
  Sleep quality will be assessed using the Pittsburgh Sleep Quality Index (PSQI). The PSQI is a validated self-report questionnaire consisting of 19 items that generate a global score ranging from 0 to 21, with higher scores indicating poorer subjective sleep quality.
  The PSQI will be administered once at baseline to characterize participants' habitual sleep quality prior to the experimental nap protocols.
Resting Heart Rate (HR) | At baseline, prior to the first experimental session.
  Resting heart rate will be measured in beats per minute (bpm) under standardized resting conditions.
  Heart rate will be recorded following a seated rest period prior to the experimental procedures to provide a baseline physiological characteristic of the participants.
Profile of Mood States (POMS) | At baseline, prior to the first experimental session.
  Mood states will be assessed using the Profile of Mood States (POMS) questionnaire.
  The POMS evaluates multiple dimensions of mood, including tension, depression, anger, vigor, fatigue, and confusion.
  Participants will complete the questionnaire under standardized conditions to characterize baseline psychological status prior to the nap interventions.

CONTACTS AND LOCATIONS:
Overall Officials: Mertkan Öncü, MsC, Study Chair — Uludag University; Monira I. Aldhahi, PhD, Principal Investigator — Nourah bint Abdulrahman University
Locations (1):
- Inonu University, Malatya, Malatya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared. The study involves a small, homogeneous sample of adolescent athletes, and the dataset includes sensitive performance and psychophysiological measures. Sharing IPD could compromise participant confidentiality and was not included in the original informed consent.

REFERENCES:
- [Result] Eken O, Oncu M, Kurtoglu A, Bozkurt O, Turkmen M, Aldhahi MI. The Acute Effects of 25- Versus 60-Minute Naps on Agility and Vertical Jump Performance in Elite Youth Soccer Players: The Role of Individual Chronotype. Life (Basel). 2025 Mar 7;15(3):422. doi: 10.3390/life15030422. PMID 40141767

DOCUMENTS (1):
  • Study Protocol (2024-05-10): https://cdn.clinicaltrials.gov/large-docs/45/NCT07314645/Prot_000.pdf